CLINICAL TRIAL: NCT04311606
Title: Anti-VEGF Therapy for Acute Thyroid Eye Disease (AcTED Study)
Brief Title: Anti-VEGF Therapy for Acute Thyroid Eye Disease
Acronym: AcTED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Nahyoung Grace Lee, MD, Physician, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019P000939
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Eye Disease
Keywords: VEGF
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: Three groups as follows:
  Group 1: Sub-tenon's injection of saline followed by sub-tenon injection of aflibercept Group 2: Sub-tenon's injection of hyaluronidase (HA) followed by sub-tenon injection of aflibercept; and Group 3: Sub-tenon injection of HA injection alone
Who Masked: Participant, Care Provider
Masking Description: Double-masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Saline and aflibercept (Experimental): Group 1: Sub-tenon's injection of saline followed by sub-tenon injection of aflibercept
  Interventions: Drug: Sub-tenon injection of saline followed by a sub-tenon injection of aflibercept
- Hyaluronidase and aflibercept (Experimental): Group 2: Sub-tenon's injection of hyaluronidase (HA) followed by sub-tenon injection of aflibercept
  Interventions: Drug: Sub-tenon injection of hyaluronidase (HA) followed by a sub-tenon injection of aflibercept
- Hyaluronidase alone (Placebo Comparator): Group 3: Sub-tenon injection of HA injection alone
  Interventions: Drug: Sub-tenon injection of hyaluronidase (HA) alone

INTERVENTIONS:
Drug: Sub-tenon injection of saline followed by a sub-tenon injection of aflibercept — The study will randomly assign a total of eight subjects into this treatment arm to receive a sub-tenon injection of saline followed by injection of 4 mg aflibercept (total volume 1.1 ml) in the worse eye. Injections will be given three times: on day 1, day 14 and day 28. Subjects will be followed until day 90.
  Other Names: Group 1
  Arms: Saline and aflibercept
Drug: Sub-tenon injection of hyaluronidase (HA) followed by a sub-tenon injection of aflibercept — The study will randomly assign a total of eight subjects into this treatment arm to receive a sub-tenon injection of hyaluronidase (HA) followed by injection of 4 mg aflibercept (total volume 1.1 ml) in the worse eye. Injections will be given three times: on day 1, day 14 and day 28. Subjects will be followed until day 90.
  Other Names: Group 2
  Arms: Hyaluronidase and aflibercept
Drug: Sub-tenon injection of hyaluronidase (HA) alone — The study will randomly assign a total of eight subjects into this treatment arm to receive a sub-tenon injection of hyaluronidase (HA) injection alone (total volume 1.1 ml) in the worse eye. Injections will be given three times: on day 1, day 14 and day 28. Subjects will be followed until day 90.
  Other Names: Group 3
  Arms: Hyaluronidase alone

SUMMARY:
The primary objective of this clinical trial is to assess the safety and tolerability of sub-tenon aflibercept in combination with either saline or hyaluronidase (HA) in patients with acute Thyroid Eye Disease (TED) as assessed by the incidence and severity of adverse events from baseline to day 45.

Participants will undergo clinical examinations and receive three injections of aflibercept with saline, aflibercept with hyaluronidase, or hyaluronidase.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum of 18 years-old
2. Active Thyroid Eye Disease
3. Clinical Activity Score (CAS) between 3 and 5, inclusive
4. Phakic and pseudophakic eyes are allowed in the study.
5. Willing and able to provide written informed consent after the nature of the study has been explained, and prior to any research-related procedures
6. Willing and able to comply with clinic visits and study-related procedures
7. Only one eye will be enrolled. The worse eye (demonstrating any of these features:

worse HVF results, worse restricted motility, worse visual acuity, worse edema, worse proptosis, worse eyelid retraction) will be enrolled. If both eyes are equivalent, we will enroll the non-dominant eye.

Exclusion Criteria:

1. History of orbital, strabismus, or eyelid surgery or orbital radiation
2. Optic neuropathy or other vision-threatening signs
3. Patients currently on systemic or topical steroids. If they received steroids in the past, they would require a 6 week washout period and the cumulative dose of steroids must be less than 1 gram of methylprednisolone (or equivalent). During the washout period we will contact patients by phone weekly to monitor their safety and address any concerns they may have related to no longer taking steroids .
4. Patients who have taken teprotumumab (Tepezza.)
5. Patients who have received intraocular anti-VEGF medications within 1 year of screening
6. Patients who have a history of receiving systemic anti-VEGF
7. Presence of other retinal vascular diseases (diabetic retinopathy, vein occlusion) that could affect the VEGF levels within the eye
8. History of stroke or prior myocardial infarction
9. Known hypersensitivity to aflibercept
10. Infectious conjunctivitis, keratitis, or endophthalmitis of either eye
11. Presence of a glaucoma shunting or filtration device that is subconjunctival
12. Previous participation in any studies of investigational drugs within 1 month preceding Day 0
13. Any clinically significant acute or chronic medical condition that would preclude participation in a clinical study
14. Pregnant or breast-feeding women
15. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)
16. History of hyaluronidase (HA) injection after the diagnosis of thyroid eye disease
17. Taking part in other research studies in the past 12 months that have involved radiation exposure
18. Participated in other research studies in the past 12 months that required radiologic imaging (particularly CT scans and not MRIs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: Safety | 45 days
  To assess the safety and tolerability of sub-tenon aflibercept in combination with either saline or hyaluronidase (HA) in patients with acute Thyroid Eye Disease (TED) as assessed by the incidence and severity of adverse events

SECONDARY OUTCOMES:
Secondary Outcome: Safety | Baseline to day 90
  To assess the safety and tolerability of sub-tenon aflibercept in combination with either saline or hyaluronidase (HA) in patients with acute Thyroid Eye Disease (TED) as assessed by the incidence and severity of adverse events
Secondary Outcome: Change in Clinical Activity | 1-90 days
  Change in clinical activity as measured by a 2 point decrease on the clinical activity score (CAS)
Secondary Outcome: Change in Ocular Muscle | 1-90 days
  Change in extra ocular muscle diameter as measured by computed tomography (CT) scan
Secondary Outcome: Change in Proptosis measured by exophthalmometry | 1-90 days
  Change in proptosis as measured by Hertel exophthalmometry
Secondary Outcome: Change in Proptosis by CT scan | 1-90 days
  Change in proptosis as measured by CT scan
Secondary Outcome: Change in Ocular Alignment | 1-90 days
  Change in degree of ocular misalignment during physical exam
Secondary Outcome: Change in Ocular Motility | 1-90 days
  Change in limitation in ocular motility as measured with physical examination
Secondary Outcome: Change in Vision measured by ETDRS BCVA | 1-90 days
  Change in vision as measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA)
Secondary Outcome: Change in Vision measured by Ishihara color test | 1-90 days
  Change in vision as measured by Ishihara color test
Secondary Outcome: Change in Visual Function | 1-90 days
  Change in visual function as determined by automated Humphrey visual field
Secondary Outcome: Change in Pain/Discomfort Reported by Subjects | 1-90 days
  Change in subjective score of pain/discomfort based upon patient Graves' Ophthalmopathy Quality of Life (GO-QOL) questionnaire
Secondary Outcome: Change in Eyelid Retraction/Position | 1-90 days
  Change in eyelid retraction/position as measured by the mm of inferior and superior scleral show on physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Nahoung Grace Lee, MD, Principal Investigator — Investigator
Locations (1):
- Mass Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant Data will be shared at end of study, after the last participant has had his or her last visit.
Supporting Information: Study Protocol, SAP
Time Frame: January 2026
Access Criteria: Email Request to PI

REFERENCES:
- [Background] Wong LL, Lee NG, Amarnani D, Choi CJ, Bielenberg DR, Freitag SK, D'Amore PA, Kim LA. Orbital Angiogenesis and Lymphangiogenesis in Thyroid Eye Disease: An Analysis of Vascular Growth Factors with Clinical Correlation. Ophthalmology. 2016 Sep;123(9):2028-36. doi: 10.1016/j.ophtha.2016.05.052. Epub 2016 Jul 14. PMID 27423310
- [Background] Smith TJ, Kahaly GJ, Ezra DG, Fleming JC, Dailey RA, Tang RA, Harris GJ, Antonelli A, Salvi M, Goldberg RA, Gigantelli JW, Couch SM, Shriver EM, Hayek BR, Hink EM, Woodward RM, Gabriel K, Magni G, Douglas RS. Teprotumumab for Thyroid-Associated Ophthalmopathy. N Engl J Med. 2017 May 4;376(18):1748-1761. doi: 10.1056/NEJMoa1614949. PMID 28467880
- [Background] Min L, Vaidya A, Becker C. Thyroid autoimmunity and ophthalmopathy related to melanoma biological therapy. Eur J Endocrinol. 2011 Feb;164(2):303-7. doi: 10.1530/EJE-10-0833. Epub 2010 Nov 18. PMID 21088057
- [Background] Kajdaniuk D, Marek B, Niedziolka-Zielonka D, Foltyn W, Nowak M, Sieminska L, Borgiel-Marek H, Glogowska-Szelag J, Ostrowska Z, Drozdz L, Kos-Kudla B. Transforming growth factor beta1 (TGFbeta1) and vascular endothelial growth factor (VEGF) in the blood of healthy people and patients with Graves' orbitopathy--a new mechanism of glucocorticoids action? Endokrynol Pol. 2014;65(5):348-56. doi: 10.5603/EP.2014.0048. PMID 25301484
- [Background] Bock F, Onderka J, Dietrich T, Bachmann B, Kruse FE, Paschke M, Zahn G, Cursiefen C. Bevacizumab as a potent inhibitor of inflammatory corneal angiogenesis and lymphangiogenesis. Invest Ophthalmol Vis Sci. 2007 Jun;48(6):2545-52. doi: 10.1167/iovs.06-0570. PMID 17525183
- [Background] Mourits MP, Koornneef L, Wiersinga WM, Prummel MF, Berghout A, van der Gaag R. Clinical criteria for the assessment of disease activity in Graves' ophthalmopathy: a novel approach. Br J Ophthalmol. 1989 Aug;73(8):639-44. doi: 10.1136/bjo.73.8.639. PMID 2765444
- [Background] Nagy JA, Vasile E, Feng D, Sundberg C, Brown LF, Detmar MJ, Lawitts JA, Benjamin L, Tan X, Manseau EJ, Dvorak AM, Dvorak HF. Vascular permeability factor/vascular endothelial growth factor induces lymphangiogenesis as well as angiogenesis. J Exp Med. 2002 Dec 2;196(11):1497-506. doi: 10.1084/jem.20021244. PMID 12461084
- [Background] Cursiefen C, Maruyama K, Jackson DG, Streilein JW, Kruse FE. Time course of angiogenesis and lymphangiogenesis after brief corneal inflammation. Cornea. 2006 May;25(4):443-7. doi: 10.1097/01.ico.0000183485.85636.ff. PMID 16670483